CLINICAL TRIAL: NCT02826681
Title: Randomized, Placebo-controlled Trial of Ferric Carboxymaltose in Restless Legs Syndrome Patients With Iron-deficiency Anemia
Brief Title: Randomized, Placebo-controlled Trial of Ferric Carboxymaltose in RLS Patients With Iron-deficiency Anemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1VIT15042
Record Dates: First submitted 2016-06-30; First posted 2016-07-11 (Estimated); Results first posted 2022-09-14 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2022-08

CONDITIONS: Restless Legs Syndrome (RLS)
MeSH Terms: conditions — Restless Legs Syndrome | interventions — ferric carboxymaltose; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Injectafer (Active Comparator): 750 mg undiluted slow IVpush (100 mg/minute) of Injectafer® (Ferric Carboxymaltose - FCM)
  Interventions: Drug: Injectafer® (Ferric Carboxymaltose - FCM)
- Normal Saline (Placebo Comparator): Placebo (15 ml of Normal Saline [NS]) IV push at 2 ml/minute on Day 0 and 7.
  Interventions: Drug: Placebo (Normal Saline)

INTERVENTIONS:
Drug: Injectafer® (Ferric Carboxymaltose - FCM) — Intravenous Iron
  Other Names: Ferinject®; Iroprem®; Renegy®
  Arms: Injectafer
Drug: Placebo (Normal Saline) — Normal Saline Solution
  Other Names: Normal Saline
  Arms: Normal Saline

SUMMARY:
Treatment Phase I and II Primary Objective: To evaluate the efficacy and safety of FCM (750 mg dose x 2) for treatment of Restless Legs Syndrome (RLS) in patients with iron-deficiency anemia (IDA).

Long-Term Extension Phase III Primary Objective: To evaluate the duration of effect of prior FCM treatment and to determine the effectiveness of further iron repletion with FCM when RLS symptoms worsen or reoccur.

DETAILED DESCRIPTION:
This will be a Phase II, randomized, placebo-controlled study. All subjects who meet the inclusion criteria, with no exclusion criteria, will qualify to enter the Screening Phase. The study will enroll 70 eligible subjects to receive blinded study drug in Treatment Phase I. All eligible subjects will be randomized in a 1:1 ratio to receive a blinded dose of either FCM 750 mg undiluted slow intravenous (IV) push at 100 mg/minute or a Placebo (15 ml of Normal Saline [NS]) IV push at 2 ml/minute on Day 0 and 7.

A subject will be defined at Day 42 as a Responder if the International Restless Legs Syndrome Severity Scale (IRLSS) score is ≤10 or if the IRLSS score is >10 with a Clinical Global Impression-Improvement (CGI-I) score of much or very much improvement and the subject does not request further treatment for RLS. A subject will be defined as a treatment Non-Responder if neither of these criteria are met.

Non-Responders who do not meet the laboratory criteria for additional dosing will be discontinued from the study and treated for RLS as deemed appropriate by the referring physician. Subjects who are Non-Responders at the end of Treatment Phase I and met the necessary laboratory criteria (ferritin <300 ng/mL and a TSAT <45%) will consented for enrollment in Treatment Phase II of the study. These subjects will receive the first of two unblinded doses of FCM (undiluted slow IV push 750 mg 100 mg/minute) on Day 0 of Phase II, which will occur within 7 days of the completing Treatment Phase I visit. The subjects will then receive the second dose of FCM (undiluted slow IV push 750 mg 100 mg/minute) on Day 7. All treated subjects will have blood samples taken for hematology, chemistries and iron indices on Day 14. Treatment efficacy (IRLSS score), medication review and adverse events assessment by phone will be done on Day 28. All subjects will return to the clinic on Day 42 for end of study assessments. Subjects completing Treatment Phase II will be re-evaluated on Day 42 and defined as either a Responder or Non-Responder, using the same criteria described above. Subjects deemed as treatment Non-Responders will be discontinued from the study after final assessments are complete.

Subjects who are evaluated on Day 42 (Week 6) as Responders from either Treatment Phase I or Treatment Phase II will continue through into the 46-Week, Long-Term Extension Phase III of the study, and be monitored and assessed by phone for RLS symptoms (IRLSS and Hopkins RLS-Sleep Quality Questionnaire [HRSQ]) and adverse events on (approximately every 9 weeks) Weeks 15, 25, 34, 43 and 52 (final follow-up visit). During Phase III subjects may receive additional unblinded treatments with FCM if at any time the subject reports worsening of RLS symptoms (an increase >4 points on the IRLSS compared to the last evaluation captured for that subject) and laboratory criteria are met (ferritin <300 ng/mL and a TSAT <45%). Subjects will receive a single FCM 750 mg undiluted slow IV push at 100 mg/minute. See section 6.6 for dosing and assessment outline. No additional treatment will be allowed after the Week 46. A final face-to-face study visit will occur on Week 52 (approximately 365 days since initial Day 0 Treatment). If a clinic visit is not possible, final evaluation will be completed by phone.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject ≥18 years of age who is able to give informed consent.
2. Confirmed diagnosis of RLS based on the Cambridge-Hopkins Diagnostic Questionnaire (CHDQ) and the Hopkins-Hening Telephone Diagnostic Interview (HDTI).
3. IRLSS score ≥15 plus RLS symptoms for at least 3 months and currently occurring ≥2 nights per week.
4. Iron-deficiency anemia defined as an Hgb <12 g/dl with a ferritin <20 ng/mL, or ferritin <100 when TSAT is <18%.
5. Subjects on sleep medication must be on a stable dose for at least 6 months prior screening.
6. Subjects at risk for pregnancy must have a negative pregnancy test at screening and be practicing an acceptable form of birth control, have had a hysterectomy or tubal ligation, or otherwise be incapable of pregnancy, or have practiced any of the following methods of contraception for at least one month prior to study entry: hormonal contraceptives, spermicide with barrier, intrauterine device, or partner sterility.

Exclusion Criteria:

1. Disorders that require treatment with the same medications used for RLS include:

   peripheral neuropathy and neurodegenerative disorders (i.e. Parkinson's disease or dementia).
2. Current (past 4 weeks) use of drugs that may cause or treat RLS, e.g. opioids, calcium channel alpha-2-delta ligands, anti-depressants, dopaminergic agonist or antagonists, or centrally-acting antihistamines.
3. Any medical conditions contraindicated to MRI.
4. Abnormal MRI at baseline that would confound the outcome measures.
5. Secondary RLS due to neurological conditions or head trauma.
6. History of hemochromatosis, hemosiderosis, other iron storage disorders or iron metabolism disorders.
7. Women with clinically significant uterine bleeding (>200 cc blood loss) during the six months prior to screening.
8. Liver transaminases (AST or ALT) greater than two times the upper limit of normal (ULN).
9. Known positive Hepatitis B antigen (HBs Ag), unless positive test can be attributed to receipt of Hepatitis B vaccination in childhood or Hepatitis C viral antibody (HCV) with evidence of active hepatitis (i.e., AST/ALT greater than two times the ULN).
10. Known positive HIV-1 or HIV-2 antibodies (anti-HIV).
11. Active acute or known chronic infections.
12. Rheumatoid arthritis with symptoms or signs of active inflammation.
13. Pregnant and lactating women.
14. Known hypersensitivity reaction to any component of Injectafer® (ferric carboxymaltose).
15. Previously randomized to Injectafer® (FCM or VIT-45) in a clinical trial.
16. Previous IV iron treatment for RLS.
17. Parenteral iron, erythropoiesis stimulating agent use or blood transfusion within six weeks prior to the screening visit.
18. Planned elective surgery during the study year.
19. Chronic alcohol or drug abuse within the past six months.
20. Any other pre-existing laboratory abnormality, medical condition, or disease that, in the opinion of Investigator, may cause the subject to be unsuitable for the study or place the subject at potential risk from being in the study, e.g. a malignancy, uncontrolled hypertension, unstable ischemic heart disease, or uncontrolled diabetes mellitus.
21. Subject is unwilling or has conditions that would prohibit them from complying with the study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2021-09-04 (Actual); Study Completion 2022-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Khechen, MD, Study Director — American Regent
Locations (8):
- United States (8):
  - Synergy San Diego, Lemon Grove, California
  - Alliance for Multispeciality Research, Fort Myers, Florida
  - CNS Healthcare, Orlando, Florida
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Boston Neuro Research, South Dartmouth, Massachusetts
  - Neurology Center of Las Vegas, Las Vegas, Nevada
  - Clinical Trial Network, Houston, Texas
  - The Polyclinic, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Monitored and assessed by phone for RLS symptoms (IRLSS and Hopkins RLS-Sleep Quality Questionnaire [HRSQ]) and TEAEs every 9 weeks ~at Weeks 15, 25, 34, 43 and 52.
  Subjects could have received additional unblinded treatments with FCM if at any time the subject reported worsening of RLS symptoms and laboratory criteria were met. No additional treatment was allowed after Week 46. final clinic visit occurred on Week 52. A clinic visit was not possible, final evaluation was completed by phone.
Period: Overall Study
Arm/Group | Injectafer | Normal Saline
Started | 35 | 35
Completed | 12 | 13
Not Completed | 23 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Injectafer | Normal Saline | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 13 | 25
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (11.46) | 44.3 (10.34) | 42.3 (10.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 25
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 9 | 16
  White | 5 | 4 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 13 | 25

OUTCOME MEASURES:

1. Primary Outcome: Treatment Phase I: IRLSS Score Change
Description: IRLSS (International Restless Legs Syndrome Severity Scale) score change from baseline to Day 42 with comparison between FCM (Ferric Carboxymaltose) vs. Placebo.
Time Frame: Baseline to Day 42
Population: Participants who were rated as much or very much improved with the CGI-I on Day 42 with comparison between Injectafer® and Placebo. CGP-I is a 7-point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention and rated as: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse.
Measure: Count of Participants; unit: Participants
Arm/Group | Injectafer | Normal Saline
Number analyzed (Participants) | 12 | 12
Participants | 12 | 12

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Injectafer | Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-04-25): https://cdn.clinicaltrials.gov/large-docs/81/NCT02826681/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-20): https://cdn.clinicaltrials.gov/large-docs/81/NCT02826681/SAP_001.pdf